CLINICAL TRIAL: NCT05970510
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ⅲ Study to Evaluate the Efficacy and Safety of Toludesvenlafaxine Hydrochloride Sustained-release Tablets in Participants With Generalized Anxiety Disorder.
Brief Title: A Study to Evaluate Efficacy and Safety of Toludesvenlafaxine Hydrochloride Sustained-release Tablets in Generalized Anxiety Disorder.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03005/CT-CHN-307
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Toludesvenlafaxine Hydrochloride Sustained-release Tablet; generalized anxiety disorder; efficacy; safety
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toludesvenlafaxine Hydrochloride Sustained-release Tablets 80 mg group (Experimental): orally once a day
  Interventions: Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablet 80mg
- Toludesvenlafaxine Hydrochloride Sustained-release Tablets 160 mg group (Experimental): orally once a day
  Interventions: Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablet 160mg
- Placebo (Sham Comparator): orally once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablet 80mg — orally once a day
  Arms: Toludesvenlafaxine Hydrochloride Sustained-release Tablets 80 mg group
Drug: Toludesvenlafaxine Hydrochloride Sustained-release Tablet 160mg — orally once a day
  Arms: Toludesvenlafaxine Hydrochloride Sustained-release Tablets 160 mg group
Drug: placebo — orally once a day
  Arms: Placebo

SUMMARY:
The study aims to evaluate the efficacy and safety of Toludesvenlafaxine Hydrochloride Sustained-release Tablets compared to placebo in adults participants with generalized anxiety disorder over a period of 8 weeks.

DETAILED DESCRIPTION:
The study consists of two periods: screening period (2 weeks) and double-blind treatment period (8 weeks). After the screening period, generalized anxiety disorder patients who satisfies the inclusion criteria are randomly assigned in the 1:1:1 ratio to receive either placebo or Toludesvenlafaxine Hydrochloride Sustained-release Tablets at two dose levels (80 ,160 mg/day) for 8 weeks. Participants are evaluated at screening, baseline visits and double-blind period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 65 years subjects;
2. Meet the Diagnostic and Statistical Manual of Manual Disorders, fifth Edition(DSM-5) criteria for Generalized Anxiety Disorder;
3. Have a Hamilton Anxiety(HAMA) Rating Scale total score ≥21 points at screening and baseline;
4. Have a Hamilton Anxiety(HAMA) Rating Scale score ≥2 points on both item 1(anxious mood) and item 2(tension) at screening and baseline;
5. Have a clinical Global Impression -severity illness (CGI-S) score≥4 points at screening and baseline.

Exclusion Criteria:

1. Meet the diagnostic criteria for other psychotic disorders(defined by DSM-5, except for GAD), including major depression disorder within 6 months prior to screening , presence or history of Schizophrenia Spectrum and Other Psychotic Disorders, Bipolar and Related Disorders, Obsessive-Compulsive and related Disorders, post-traumatic stress disorder, anorexia nervosa or bulimia and personality disorder;
2. Meet the diagnostic criteria for substance or alcohol abuse (defined by DSM-5, except for nicotine or caffeine) within 6 months prior to screening;
3. Have anxious symtoms secondary to other physical illnesses or mental illnesses and anxious induced by psychoactive substance;
4. Withdrawal psychotropic drugs within 5 half-lives (at least 2 weeks for monoamine oxidase inhibitors, at least 1 month for fluoxetine, and at least 2 weeks for benzodiazepines or barbiturates) prior to randomization;
5. Have received psychosurgery or physical therapy for psychiatric illness (such as transcranial magnetic stimulation) within 3 months prior to screening;
6. Have received systematic psychotherapy or other non-drug therapies for psychiatric disorders (such as acupuncture or light therapy) within 6 weeks prior to screening;
7. Concomitant with serious and unstable illness, including cardiovascular, hepatic, renal, hematological, endocrine illness, malignant tumors and other physical illness;
8. Have a history of seizures (except for seizures caused by febrile convulsions in childhood);
9. Have a history of gastrointestinal disease or surgery known to interfere with investigation product absorption or excretion;
10. Known or suspected allergic or severe reaction to investigation product or inactive ingredients; or allergic to venlafaxine or desvenlafaxine; or allergic constitution (defined as allergic to two or more drugs or food) and unfit to participate judged by investigator;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Hamilton Anxiety(HAMA) Rating Scale total score at endpoint | from baseline to week 8
  The HAMA Scale consist of 14 items that include psychic, somatic, and behavioral symptoms associated with anxiety. Each items is rated on a 5-point scale of 0(not present) to 4(very severe) so that scores may range from 0 to 56, with high scores indicating greater illness severity.

SECONDARY OUTCOMES:
Change from baseline in the Hamilton Anxiety(HAMA) Rating Scale psychic factor score (Items 1~6 and Item 14) at endpoint | from baseline to week 8
  The psychic factor score is the sum of items 1-6 and items 14(including items such as anxious mood, tension, fear, insomnia, and behavioral symptoms).Each items is rated on a 5-point scale of 0(not present) to 4(very severe) so that scores may range from 0 to 28, with high scores indicating greater illness severity.
Change from baseline in the Hamilton Anxiety(HAMA) Rating Scale somatic factor score (Items 7~13) at endpoint | from baseline to week 8
  The somatic factor score is the sum of items 7-13(including items such as cardiovascular, respiratory, and gastrointestinal symptoms).Each items is rated on a 5-point scale of 0(not present) to 4(very severe) so that scores may range from 0 to 28, with high scores indicating greater illness severity.
Change from baseline in the Hamilton Anxiety(HAMA) Rating Scale item 1（Anxious mood）Score at endpoint | from baseline to week 8
  The item is rated on a 5-point scale of 0(not present) to 4(very severe) so that score may range from 0 to 4, with high scores indicating greater illness severity.
Change from baseline in the Hamilton Anxiety(HAMA) Rating Scale item 2（Tension）Score at endpoint | from baseline to week 8
  The item is rated on a 5-point scale of 0(not present) to 4(very severe) so that score may range from 0 to 4, with high scores indicating greater illness severity.
Percentage of participants with response at endpoint | from baseline to week 8
  Response was defined as a≥50% reduction from baseline to endpoint in the HAMA total score.
Percentage of participants with remission at endpoint | from baseline to week 8
  Remission was defined as a HAMA total score ≤7 points at endpoint
Clinical Global Impression Scale - improvement (CGI-I) score at endpoint | from baseline to week 8
  The CGI-I scale measures the participant's improvement (or worsening) as assessed by the investigator relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Change from baseline in Clinical Global Impression Scale - severity (CGI-S) score at endpoint | from baseline to week 8
  The CGI-S scale is a 7-point scale to rate the severity of the patient's illness. Patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Change from baseline in the Sheehan Disability Scale(SDS) score at endpoint | from baseline to week 8
  The SDS scale consists of 3 items evaluating impairment in work/school， social life/leisure activities, and family life/home responsibilities. Each item is scored on a scale of 0(unimpaired) to 10(highly impaired).
Change from baseline in the Pittsburgh Sleep Quality Index (PSQI) score at endpoint | from baseline to week 8
  The scale consists of 3 items evaluating impairment in work/school， social life/leisure activities, and family life/home responsibilities. Each item is scored on a scale of 0(unimpaired) to 10(highly impaired).
Incidence and severity of adverse effects (AEs) | from baseline to week 8
Change from baseline in the Columbia Suicide severity Rating Scale (C-SSRS) score at endpoint | from baseline to week 8
  The C-SSRS captured the occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation: a "yes" answer to any 1 of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation. Suicidal behavior: a "yes" answer to any 1 of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Hongyan, Principal Investigator — Peking University Sixth Hospital
Locations (1):
- Peking University Sixth Hospital, Beijing, China